CLINICAL TRIAL: NCT03858062
Title: Algorithm to Control Postprandial, Post Exercise and Night Glucose Excursions in a Portable Closed Loop Format, APPEL 5
Brief Title: Algorithm to Control Postprandial, Post Exercise and Night Glucose Excursions in a Portable Closed Loop Format,
Acronym: APPEL5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J.H. DeVries (Other)
Collaborators: Rijnstate Hospital (Other); Inreda Diabetic B.V. (Industry)
Responsible Party: Sponsor-Investigator, J.H. DeVries, Endocrinologist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL55693.018.15
Record Dates: First submitted 2019-02-21; First posted 2019-02-28 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Artificial pancreas; Glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open loop (Active Comparator): 14 days patient-managed Insulin pump therapy (with or without glucose sensor) with blinded continuous glucose monitoring
  Interventions: Device: Insulin pump therapy (with or without glucose sensor)
- Closed loop (Experimental): 4-6 training + 14 days automated blood glucose control with the Artificial pancreas (Inreda Diabetic)
  Interventions: Device: Artificial pancreas (Inreda Diabetic)

INTERVENTIONS:
Device: Insulin pump therapy (with or without glucose sensor) — Patients' own insulin pump with fast-acting insulin analog and optionally with own glucose sensor
  Other Names: Continuous subcutaneous insulin infusion (CSII); Sensor augmented pump therapy (SAP)
  Arms: Open loop
Device: Artificial pancreas (Inreda Diabetic) — Bi-hormonal reactive closed loop system without mealtime announcement
  Other Names: Closed loop therapy
  Arms: Closed loop

SUMMARY:
In previous studies, the investigators tested the feasibility of a bi-hormonal reactive closed loop system without mealtime announcement. This system for automated control of blood glucose in patients with type 1 diabetes was tested in the clinical research center (APPEL 1 and 2) as well as at the home of the patients (APPEL 3 and 4). After the APPEL 4 study some improvements have been made to the miniaturized prototype to allow patients to operate the system independently and additional risk control measures were included. The main objective of this study is to assess the efficacy of this improved closed loop system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus type 1;
* Treated with SAP or CSII for a minimum of 6 months;
* Willing and able to sign informed consent.

Exclusion Criteria:

* Impaired awareness of hypoglycemia (score ≥ 4) according to Gold and/or Clarke questionnaire;
* BMI > 35 kg/m2;
* HbA1c > 97 mmol/mol (=11.0 %);
* Use of heparin, coumarin derivatives or oral corticosteroids;
* Use of acetaminophen during the open loop or closed loop period, as this may influence the sensor glucose measurements;
* Limited ability to see, and to hear or feel alarm signals of the closed loop system;
* Skin condition prohibiting needle insertion;
* Pregnancy and/or breastfeeding;
* Living alone during the night during the closed loop period (the patient may ask someone to stay over temporarily);
* Expected poor connectivity with internet regarding 24/7 tele monitoring;
* Any condition that the local investigator feels would have interfere with trial participation or the evaluation of the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Time in target | Week 1-2
  Proportion of time spent in the target range (3.9-10 mmol/l)

SECONDARY OUTCOMES:
Time in hypoglycemia 1 | Week 1-2 / Week 1 / Week 2
  Proportion of time spent in hypoglycemia (<3.9 mmol/l)
Time in hypoglycemia 2 | Week 1-2 / Week 1 / Week 2
  Proportion of time spent in hypoglycemia (<3.3 mmol/l)
Time in hyperglycemia 1 | Week 1-2 / Week 1 / Week 2
  Proportion of time spent in hyperglycemia (>10 mmol/l)
Time in hyperglycemia 2 | Week 1-2 / Week 1 / Week 2
  Proportion of time spent in hyperglycemia (>13.9 mmol/l)
Hypoglycemic events | Week 1-2 / Week 1 / Week 2
  Number of carbohydrate-treated hypoglycemic events
Mean or median glucose | Week 1-2 / Week 1 / Week 2
  Mean or median sensor glucose concentration
Mean or median day glucose | Day time: Week 1-2 / Week 1 / Week 2
  Mean or median sensor glucose concentration
Mean or median night glucose | Night time: Week 1-2 / Week 1 / Week 2
  Mean or median sensor glucose concentration
Mean or median postprandial glucose | Postprandial: Week 1-2 / Week 1 / Week 2
  Mean or median sensor glucose concentration
Glycemic variability 1 | Week 1-2 / Week 1 / Week 2
  Interquartile range (IQR)
Glycemic variability 2 | Week 1-2 / Week 1 / Week 2
  Coefficient of variation (CV)
Glycemic variability 3 | Week 1-2 / Week 1 / Week 2
  Low blood glucose index (LBGI)
Glycemic variability 4 | Week 1-2 / Week 1 / Week 2
  High blood glucose index (HBGI)
Glycemic variability 5 | Week 1-2 / Week 1 / Week 2
  Blood glucose risk index (BGRI)
Time in target | Week 1 / Week 2
  Proportion of time spent in the target range (3.9-10 mmol/l)
PAID: Problem Areas In Diabetes questionnaire | Baseline / End week 2
  Total score; Scale 0 (no problems) to 80 (big problems)
EQ5D: EuroQol 5 Dimensions questionnaire | Baseline / End week 2
  Quality of life measure; Scale 1 ("no problem) to 5 ("extreme problems")
DTSQ-status: Diabetes Treatment Satisfaction Questionnaire | Baseline / End week 2
  Total score: Scale 0 (negative) to 36 (positive)
DTSQ-change: Diabetes Treatment Satisfaction Questionnaire | End week 2
  Change in DTSQ; Total score: Scale -18 (negative) to 18 (positive)
Algorithm active time | Week 1-2 (closed loop only)
  Percentage of time that the closed loop algorithm is active
Usability score | End week 2 (closed loop only)
  Questionnaire: Mobile Phone Usability Questionnaire (MPUQ); Total score: Scale 62 (low level of usability) to 310 (higher level of usability)
Glucose measurement performance | Day 3, 4 or 5 of the training period prior to the closed loop
  MARD

OTHER OUTCOMES:
Demographic variables | Baseline
Weight | Baseline
Length | Baseline
HbA1c plasma concentration | Baseline
Meals | Week 1-2
  Carbohydrate intake
Physical activity 1 | Week 1-2
  Number of exercise moments per intensity category ("light", "moderate", "heavy'"
  )
Physical activity 2 | Week 1-2
  Duration of exercise moments per intensity category ("light", "moderate", "heavy'"
  )
Physical activity 3 | Week 1-2
  Total number of exercise moments
Physical activity 4 | Week 1-2
  Total duration of exercise moments
Insulin dose | Week 1-2
  Daily average
Glucagon dose | Week 1-2
  Daily average

CONTACTS AND LOCATIONS:
Overall Officials: J.H. DeVries, MD PhD, Principal Investigator — Academisch Medisch Centrum, Universiteit van Amsterdam
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Academic Medical Center, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Bon AC, Luijf YM, Koebrugge R, Koops R, Hoekstra JB, DeVries JH. Feasibility of a portable bihormonal closed-loop system to control glucose excursions at home under free-living conditions for 48 hours. Diabetes Technol Ther. 2014 Mar;16(3):131-6. doi: 10.1089/dia.2013.0166. Epub 2013 Nov 13. PMID 24224750
- [Background] Blauw H, van Bon AC, Koops R, DeVries JH; , on behalf of the PCDIAB consortium. Performance and safety of an integrated bihormonal artificial pancreas for fully automated glucose control at home. Diabetes Obes Metab. 2016 Jul;18(7):671-7. doi: 10.1111/dom.12663. Epub 2016 Apr 25. PMID 26996542
- [Derived] Blauw H, Onvlee AJ, Klaassen M, van Bon AC, DeVries JH. Fully Closed Loop Glucose Control With a Bihormonal Artificial Pancreas in Adults With Type 1 Diabetes: An Outpatient, Randomized, Crossover Trial. Diabetes Care. 2021 Mar;44(3):836-838. doi: 10.2337/dc20-2106. Epub 2021 Jan 4. PMID 33397767